CLINICAL TRIAL: NCT03422757
Title: A Double Blind, Crossover Study to Evaluate Safety and Efficacy of an Adaptive Deep Brain Stimulation Closed-loop Method Compared With Conventional Deep Brain Stimulation in Patients With Parkinson's Disease
Brief Title: Safety and Efficacy of Adaptive DBS Vs Conventional DBS in Patients With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: Newronika (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NWK_aDBSext_01_2017
Record Dates: First submitted 2017-12-15; First posted 2018-02-06 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adaptive DBS (Experimental): adaptive Deep Brain Stimulation, by AlphaDBSvext.
  Interventions: Device: adaptive Deep Brain Stimulation
- conventional DBS (Active Comparator): conventional Deep Brain Stimulation, by AlphaDBSvext.
  Interventions: Device: conventional Deep Brain Stimulation

INTERVENTIONS:
Device: adaptive Deep Brain Stimulation — The investigational medical device ("AlphaDBSvext") is a portable, external, dual mode stimulator that can deliver adaptive DBS or conventional DBS for the treatment of PD.
  In the adaptive mode, the device records Local Field Potential activity from the implanted DBS electrode and simultaneously delivers stimulation through the same electrode based on the recorded signal.
  Arms: adaptive DBS
Device: conventional Deep Brain Stimulation — The same investigational medical device ("AlphaDBSvext") is used to deliver conventional DBS for the treatment of PD. In the conventional mode it delivers constant stimulation.
  Arms: conventional DBS

SUMMARY:
This is an exploratory study to preliminary assess safety and efficacy of an adaptive Deep Brain Stimulation (DBS) closed-loop method in patients with PD.

The study has been designed as a double blind randomized crossover trial that uses conventional DBS as a concurrent control in PD patients in need of Implantable Pulse Generator (IPG) replacement.

DETAILED DESCRIPTION:
PD patients in need of IPG replacement will be screened to identify the ones eligible for enrollment.

Randomized patients will undergo 2 days of experimental sessions (i.e. one per each type of stimulation mode, cDBS and aDBS), in a well-controlled environment (i.e. during hospitalization). During each experimental session experienced neurologists will collect information on safety and efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD;
* DBS implant since at least 3 years and in need of battery replacement, defined by battery level <25%;
* Patients must be able to sign the informed consent document to participate in the clinical trial;
* Patients with a suboptimal response to DBS treatment.

Exclusion Criteria:

* Patients with severe cognitive decline (MMSE <25);
* Patients with major psychiatric issues;
* Patients with any medical condition potentially interfering with DBS battery replacement surgery;
* Patients that cannot tolerate an interruption of DBS stimulation;
* Patients taking only one levodopa dose per day;
* Patients with no LFPs recorded from any contacts pair, during intraoperatory IPG replacement procedure;
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Total Electrical Energy Delivered (TEED) to the patient | One day.
  Difference in the TEED delivered to the patient in adaptive DBS versus conventional DBS mode.

SECONDARY OUTCOMES:
Incidence of device related Adverse Events (safety and tolerability) | One day.
  Number of device relate Adverse Events or abnormal vital signs.
Unified Parkinson's Disease Rating Scale (UPDRS) part III | One day.
  Evaluation of motor symptoms through (UPDRS) part III, motor examination. The total score is computed from scores obtained on 18 items (0 best condition-4 worst condition), some considering multiple body parts.
Unified Dyskinesia Rating Scale (UDysRS) | One day.
  Evaluation of dyskinesia through repeated clinical assessments (using UDysRS).

OTHER OUTCOMES:
Time "off" | One day.
  Evaluation of time "off" through patient diary.
DBS Impairment Scale (DBS-IS) | One day.
  Self assessment through questionnaire.
Local field potentials (LFP) during gait analysis | Four hours.
  Evaluation of LFP recording from DBS electrodes during gait analysis.
Local field potentials (LFP) during speech analysis | Four hours.
  Evaluation of LFP recording from DBS electrodes during speech analysis.
Local field potentials (LFP) during sleep analysis | One night.
  Evaluation of LFP recording from DBS electrodes during sleep analysis.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Centro Parkinson e Disturbi del Movimento ASST G.Pini- CTO, Milan
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, Pavia